CLINICAL TRIAL: NCT03209713
Title: Edtech-HPV: A Community Approach Using Education and Technology to Increase HPV Vaccination
Acronym: Edtech-HPV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-336
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Parents
Keywords: Mexican; Mexican-American; 17-336

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental Education (Active Comparator): Participants will receive parental education on HPV vaccine and the vaccine's benefits.
  Interventions: Behavioral: HPV Vaccine Education
- Parental Education + Text Messaging (Experimental): Participants will receive parental education on HPV vaccine and the vaccine's benefits plus text messaging reminder.
  Interventions: Behavioral: HPV Vaccine Education; Behavioral: Text Messaging Reminder

INTERVENTIONS:
Behavioral: HPV Vaccine Education — A one on one twenty-minute parental educational program (in-person or over the phone) providing facts about HPV, HPV-related cancers, and the HPV vaccine.
Behavioral: Text Messaging Reminder — Participants will receive a text message reminding them of their child's vaccination eligibility once a week, starting one week after participating in the education session (in-person or over the phone). All participants randomized to the text message reminder arm will receive a welcome text message from the automated web-based text messaging service, Mosio, within 72 hours from registration. One week after receiving the welcome text message, they will receive the first weekly text messages reminding them of their child's eligibility for the first dose HPV vaccine. These weekly reminders will occur until uptake of the first dose of the vaccine is reported (through self-report outcome survey completion or submission of the HPV vaccination card/child's official immunization card) or for up to 12 weeks
  Other Names: EdTech-HPV
  Arms: Parental Education + Text Messaging

SUMMARY:
This study is a two-arm randomized controlled trial, implemented to assess the effectiveness of a community-based educational program with and without a text messaging reminder system, in increasing the rate of HPV vaccination completion among children of Mexican Americans.

The investigator's have extended the duration that participants are followed in assessing their child's uptake of the HPV vaccine to coincide with the COVID-19 related clinic closures and/or allow flexibility for participants who decide to delay their child's vaccination for fear of exposure to the COVID-19 infection.

A survey will also assess the participants concerns regarding the impact COVID-19 has had in their daily life, such as financial insecurity, food access, housing insecurity and among other most common concerns during this unprecedented time. Additional navigation, referrals and interviewer notes will also be captured. Participants may be called by site or MSK staff to complete study surveys and will be informed verbally or by a mailed letter.

ELIGIBILITY:
Inclusion Criteria:

* Born in Mexico or born in U.S. but self-describes as Mexican-American
* Spanish is his or her primary language
* Has a minimum of one child between the ages of 11 and 17 who has not initiated or completed the HPV vaccine seriest (as per the age-recommended timeframe)
* Self-identifies as the child's main caregiver
* Currently owns a cell phone and uses text messaging services and is willing to accept text messages for this study
* 21 to 84 years old

Exclusion Criteria:

* Presence of a serious psychiatric or cognitive impairment likely to preclude meaningful informed consent and adherence to the protocol per the consenting professional's judgment.

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Vaccination completion assessment rate | 2 years
  Comparison rates of vaccination completion will be assessed by Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Alivio Medical Center, Chicago, Illinois
  - Research, Education and Access to Community Health (REACH), Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas at El Paso, El Paso, Texas

REFERENCES:
- [Derived] Aragones A, Zamore C, Moya EM, Cordero JI, Gany F, Bruno DM. The Impact of Restrictive Policies on Mexican Immigrant Parents and Their Children's Access to Health Care. Health Equity. 2021 Sep 14;5(1):612-618. doi: 10.1089/heq.2020.0111. eCollection 2021. PMID 34909528
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org